CLINICAL TRIAL: NCT06098300
Title: Effects of Change in Blood Pressure on Retinal Capillary Rarefaction in Patients With Arterial Hypertension - a Pilot Study
Brief Title: Effects of Change in Blood Pressure on Retinal Capillary Rarefaction in Patients With Arterial Hypertension
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Principal Investigator, Medical University of Vienna
Other Study IDs: OPHT-240323
Record Dates: First submitted 2023-09-05; First posted 2023-10-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Arterial Hypertension; Blood Pressure, High
Keywords: Retinal Capillary Rarefaction; Hypertension; Antihypertensive medication; OCT-A; Retinal oxygen extraction; Choroidal vascularity index (CVI); Ocular blood flow
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate whether in patients with initially poorly-controlled arterial hypertension, structural and functional differences in the retina and choroid remain after achieving a well-controlled blood pressure.

DETAILED DESCRIPTION:
Optical Coherence Tomography Angiography (OCT-A) is an ocular imaging technique which allows fast and non-invasive assessment of the retinal microvasculature. With the OCT-A, a reduction in capillary density in patients with arterial hypertension has been found. In animal experiments, this so called retinal capillary rarefaction could be reversed after administration of antihypertensive medication.

The main aim of the present study is to evaluate whether in patients with initially poorly-controlled hypertension, an increase in capillary density can be demonstrated, if patients achieve well-controlled blood pressure with antihypertensive medication. In addition changes in retinal oxygen metabolism and choroidal blood flow will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged ≥ 18 years
* Signed informed consent
* Apart from hypertensive retinopathy, normal ophthalmic findings
* Non-Smokers
* Patients with initially diagnosed or pre-existing mild to moderate primary arterial hypertension (systolic office blood pressure ≥ 140 mmHg and/or diastolic office blood pressure ≥ 90 mmHg)
* Planned initiation of antihypertensive medication or planned adaption of antihypertensive medication by the Department of Cardiology
* Subject agrees to perform regular blood pressure self-measurements and to document blood pressure values in a diary

Exclusion Criteria:

* Participation in a clinical trial in the three weeks preceding the study
* Blood donation in the three weeks preceding the study
* Symptoms of a clinically relevant illness in the three weeks preceding the study
* History of family history of epilepsy
* Secondary hypertension (e.g.: hyperaldosteronism, pheochromocytoma, renal artery stenosis, renal parenchymal diseases, Cushing-syndrome, Coarctatio aortae)
* History of hypertensive encephalopathy or intracerebral bleeding
* Diabetes mellitus Type 1 or Type 2
* Pregnant or breast-feeding women
* Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with initially diagnosed or pre-existing mild to moderate primary arterial hypertension (systolic office blood pressure ≥ 140 mmHg and/or diastolic office blood pressure ≥ 90 mmHg) with a planned initiation or planned adaption of antihypertensive medication by the Department of Cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in retinal vessel density after achieving blood pressure treatment target (OCT-A). | 12 weeks
  As OCT devices are able to calculate the movements of erythrocytes, retinal perfusion can be visualized with Optical Coherence Tomography Angiography. No contrast media is necessary for the representation of retinal vessels.

SECONDARY OUTCOMES:
Change in choroidal vascularity index after achieving blood pressure treatment target (EDI-OCT). | 12 weeks
  The choroid will be imaged with the enhanced-depth-imaging-OCT (EDI-OCT) (Spectralis, Heidelberg Engineering, Heidelberg, Germany). By using an automatic detection algorithm, developed by Tian et al., the choroid will be separated from the sclera and Bruch´s membrane. Afterwards, the image will be binarized using the software Fiji ImageJ. An autolocal threshold will be applied and the image will be converted into an RGB (red, green, blue) image, thereby determining the luminal area of the choroid. The choroidal vascularity index is obtained by dividing the luminal area by the total choroidal area.
Change in neurovascular coupling after achieving blood pressure treatment target (DVA). | 12 weeks
  The DVA allows for the real time measurement of retinal vessel diameters in vivo. The DVA is a commercially available system (IMEDOS, Jena, Germany) which comprises a fundus camera, a video camera, a real time monitor and a personal computer with an analyzing software for the accurate determination of retinal arterial and venous diameters. Every second a maximum of 25 readings of vessel diameter can be obtained. For this purpose the fundus is imaged onto the charge coupled device chip of the video camera. The consecutive fundus images are digitized using a frame grabber. In addition, the fundus image can be inspected on the real time monitor and, if necessary, stored on a video recorder. Evaluation of the retinal vessel diameters can either be done online or offline from the recorded video tapes.
Change in retinal oxygen saturation after achieving blood pressure treatment target (DVA). | 12 weeks
  Retinal oxygen saturation measurement is based on the image analysis by the oxygen module of the commercially available Dynamic Vessel Analyzer (DVA, Imedos, Germany). Two monochromatic fundus images are recorded by the retinal oximeter. In an image, obtained by the camera and filter assembly, the operator has to mark the vessel of interest by a mouse click. The vessel is traced automatically applying the following procedure. The vessel walls are located as photometric edges in the vicinity of the mouse cursor in the green channel image. If edges are determined, the search is continued in their proximity.
Change in ocular blood flow after achieving blood pressure treatment target (LSFG). | 12 weeks
  A commercially available LSFG (Nidek, Japan) system will be used in the present study. The LSFG device consists of a fundus camera equipped with a diode laser with a wavelength of 830 nm and a charge-coupled device. NB, the relative velocity of blood flow, is derived from the pattern of speckle contrast produced by the interference of a laser scattered by blood cells moving in the ocular fundus. Images are acquired continuously at the rate of 30 frames per seconds in a 4-second time period and stored on a personal computer. Equipped analysis software synchronizes the captured MBR images in each cardiac cycle, and averages the MBR in each heartbeat to produce a heartbeat map of the ONH and the retina/choroid.
Change in retinal oxygen extraction after achieving blood pressure treatment target. | 12 weeks
  Retinal oxygen extraction will be determined by measuring retinal blood flow (LSFG), retinal oxygen saturation (DVA) and retinal vessel diameter (DVA). For the calculation of retinal oxygen extraction, the formula of Werkmeister et al. will be used, which will be slightly modified as retinal blood flow is measured with LSFG and not with Doppler OCT.
Change in ocular perfusion pressure and arterial blood pressure after achieving blood pressure treatment target. | 12 weeks
  mOPP = 2/3 mBP- IOP Blood pressure will be measured with an automated oscillometric device
Change in retinal vessel diameter after achieving blood pressure treatment target (DVA). | 12 weeks
  Two monochromatic fundus images are recorded by the retinal oximeter. In an image, obtained by the camera and filter assembly, the operator has to mark the vessel of interest by a mouse click. The vessel is traced automatically applying the following procedure. The vessel walls are located as photometric edges in the vicinity of the mouse cursor in the green channel image. If edges are determined, the search is continued in their proximity.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Mills KT, Stefanescu A, He J. The global epidemiology of hypertension. Nat Rev Nephrol. 2020 Apr;16(4):223-237. doi: 10.1038/s41581-019-0244-2. Epub 2020 Feb 5. PMID 32024986
- [Background] Dai H, Bragazzi NL, Younis A, Zhong W, Liu X, Wu J, Grossman E. Worldwide Trends in Prevalence, Mortality, and Disability-Adjusted Life Years for Hypertensive Heart Disease From 1990 to 2017. Hypertension. 2021 Apr;77(4):1223-1233. doi: 10.1161/HYPERTENSIONAHA.120.16483. Epub 2021 Feb 15. PMID 33583201
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752
- [Background] Dziedziak J, Zaleska-Zmijewska A, Szaflik JP, Cudnoch-Jedrzejewska A. Impact of Arterial Hypertension on the Eye: A Review of the Pathogenesis, Diagnostic Methods, and Treatment of Hypertensive Retinopathy. Med Sci Monit. 2022 Jan 20;28:e935135. doi: 10.12659/MSM.935135. PMID 35046380
- [Background] Oh JS, Lee CH, Park JI, Park HK, Hwang JK. Hypertension-Mediated Organ Damage and Long-term Cardiovascular Outcomes in Asian Hypertensive Patients without Prior Cardiovascular Disease. J Korean Med Sci. 2020 Dec 14;35(48):e400. doi: 10.3346/jkms.2020.35.e400. PMID 33316856
- [Background] Unger T, Borghi C, Charchar F, Khan NA, Poulter NR, Prabhakaran D, Ramirez A, Schlaich M, Stergiou GS, Tomaszewski M, Wainford RD, Williams B, Schutte AE. 2020 International Society of Hypertension Global Hypertension Practice Guidelines. Hypertension. 2020 Jun;75(6):1334-1357. doi: 10.1161/HYPERTENSIONAHA.120.15026. Epub 2020 May 6. No abstract available. PMID 32370572
- [Background] Wong TY, Mitchell P. The eye in hypertension. Lancet. 2007 Feb 3;369(9559):425-35. doi: 10.1016/S0140-6736(07)60198-6. PMID 17276782
- [Background] Kurniawan ED, Cheung N, Cheung CY, Tay WT, Saw SM, Wong TY. Elevated blood pressure is associated with rarefaction of the retinal vasculature in children. Invest Ophthalmol Vis Sci. 2012 Jan 31;53(1):470-4. doi: 10.1167/iovs.11-8835. PMID 22205607
- [Background] Chua J, Chin CWL, Hong J, Chee ML, Le TT, Ting DSW, Wong TY, Schmetterer L. Impact of hypertension on retinal capillary microvasculature using optical coherence tomographic angiography. J Hypertens. 2019 Mar;37(3):572-580. doi: 10.1097/HJH.0000000000001916. PMID 30113530
- [Background] Jumar A, Harazny JM, Ott C, Kistner I, Friedrich S, Schmieder RE. Improvement in Retinal Capillary Rarefaction After Valsartan Treatment in Hypertensive Patients. J Clin Hypertens (Greenwich). 2016 Nov;18(11):1112-1118. doi: 10.1111/jch.12851. Epub 2016 Jun 16. PMID 27306560
- [Background] Bosch AJ, Harazny JM, Kistner I, Friedrich S, Wojtkiewicz J, Schmieder RE. Retinal capillary rarefaction in patients with untreated mild-moderate hypertension. BMC Cardiovasc Disord. 2017 Dec 21;17(1):300. doi: 10.1186/s12872-017-0732-x. PMID 29268712
- [Background] Chua J, Le TT, Tan B, Ke M, Li C, Wong DWK, Tan ACS, Lamoureux E, Wong TY, Chin CWL, Schmetterer L. Choriocapillaris microvasculature dysfunction in systemic hypertension. Sci Rep. 2021 Feb 25;11(1):4603. doi: 10.1038/s41598-021-84136-6. PMID 33633311
- [Background] Schrimpf C, Teebken OE, Wilhelmi M, Duffield JS. The role of pericyte detachment in vascular rarefaction. J Vasc Res. 2014;51(4):247-58. doi: 10.1159/000365149. Epub 2014 Sep 3. PMID 25195856
- [Background] Estato V, Obadia N, Carvalho-Tavares J, Freitas FS, Reis P, Castro-Faria Neto H, Lessa MA, Tibirica E. Blockade of the renin-angiotensin system improves cerebral microcirculatory perfusion in diabetic hypertensive rats. Microvasc Res. 2013 May;87:41-9. doi: 10.1016/j.mvr.2013.02.007. Epub 2013 Mar 1. PMID 23466285
- [Background] Sabino B, Lessa MA, Nascimento AR, Rodrigues CA, Henriques Md, Garzoni LR, Levy BI, Tibirica E. Effects of antihypertensive drugs on capillary rarefaction in spontaneously hypertensive rats: intravital microscopy and histologic analysis. J Cardiovasc Pharmacol. 2008 Apr;51(4):402-9. doi: 10.1097/FJC.0b013e3181673bc5. PMID 18427284
- [Background] Rizzoni D, Porteri E, Boari GE, De Ciuceis C, Sleiman I, Muiesan ML, Castellano M, Miclini M, Agabiti-Rosei E. Prognostic significance of small-artery structure in hypertension. Circulation. 2003 Nov 4;108(18):2230-5. doi: 10.1161/01.CIR.0000095031.51492.C5. Epub 2003 Oct 13. PMID 14557363
- [Background] Agabiti-Rosei E, Rizzoni D. Microvascular structure as a prognostically relevant endpoint. J Hypertens. 2017 May;35(5):914-921. doi: 10.1097/HJH.0000000000001259. PMID 28355167
- [Background] Chua J, Le TT, Sim YC, Chye HY, Tan B, Yao X, Wong D, Ang BWY, Toh DF, Lim H, Bryant JA, Wong TY, Chin CWL, Schmetterer L. Relationship of Quantitative Retinal Capillary Network and Myocardial Remodeling in Systemic Hypertension. J Am Heart Assoc. 2022 Mar 15;11(6):e024226. doi: 10.1161/JAHA.121.024226. Epub 2022 Mar 5. PMID 35253475
- [Background] Sun C, Ladores C, Hong J, Nguyen DQ, Chua J, Ting D, Schmetterer L, Wong TY, Cheng CY, Tan ACS. Systemic hypertension associated retinal microvascular changes can be detected with optical coherence tomography angiography. Sci Rep. 2020 Jun 12;10(1):9580. doi: 10.1038/s41598-020-66736-w. PMID 32533105
- [Background] Lee WH, Park JH, Won Y, Lee MW, Shin YI, Jo YJ, Kim JY. Retinal Microvascular Change in Hypertension as measured by Optical Coherence Tomography Angiography. Sci Rep. 2019 Jan 17;9(1):156. doi: 10.1038/s41598-018-36474-1. PMID 30655557
- [Background] Terheyden JH, Wintergerst MWM, Pizarro C, Pfau M, Turski GN, Holz FG, Finger RP. Retinal and Choroidal Capillary Perfusion Are Reduced in Hypertensive Crisis Irrespective of Retinopathy. Transl Vis Sci Technol. 2020 Jul 29;9(8):42. doi: 10.1167/tvst.9.8.42. eCollection 2020 Jul. PMID 32855888
- [Background] Frost S, Nolde JM, Chan J, Joyson A, Gregory C, Carnagarin R, Herat LY, Matthews VB, Robinson L, Vignarajan J, Prentice D, Kanagasingam Y, Schlaich MP. Retinal capillary rarefaction is associated with arterial and kidney damage in hypertension. Sci Rep. 2021 Jan 13;11(1):1001. doi: 10.1038/s41598-020-79594-3. PMID 33441624
- [Background] Antonios TF, Singer DR, Markandu ND, Mortimer PS, MacGregor GA. Structural skin capillary rarefaction in essential hypertension. Hypertension. 1999 Apr;33(4):998-1001. doi: 10.1161/01.hyp.33.4.998. PMID 10205237
- [Background] Weber T, Arbeiter K, Ardelt F, Auer J, Aufricht C, Brandt MC, Dichtl W, Ferrari J, Foger B, Henkel M, Hohenstein-Scheibenecker K, Horn S, Kautzky-Willer A, Kepplinger E, Knoflach M, Koppelstatter C, Mache C, Marschang P, Mayer G, Metzler B, Oberbauer R, Obermair F, Obermayer-Pietsch B, Perl S, Pilz S, Prischl FC, Podczeck-Schweighofer A, Rebhandl E, Rohla M, Roller-Wirnsberger R, Saely CH, Siostrzonek P, Slany J, Stoschitzky K, Waldegger S, Wenzel RR, Weiss T, Wirnsberger G, Winhofer-Stockl Y, Zweiker D, Zweiker R, Watschinger B; Osterreichische Gesellschaft fur Hypertensiologie; Osterreichische Atherosklerosegesellschaft; Osterreichische Diabetes Gesellschaft; Osterreichische Gesellschaft fur Internistische Angiologie; Osterreichische Gesellschaft fur Nephrologie; Osterreichische Kardiologische Gesellschaft; Osterreichische Gesellschaft fur Neurologie; Osterreichische Schlaganfall-Gesellschaft; Osterr. Gesellschaft fur Allgemeinmedizin; Osterr. Gesellschaft fur Geriatrie; Osterreichische Gesellschaft fur Endokrinologie und Stoffwechsel; Osterreichische Gesellschaft fur Innere Medizin; Osterreichische Gesellschaft fur Kinder- und Jugendheilkunde. [Austrian Consensus on High Blood Pressure 2019]. Wien Klin Wochenschr. 2019 Nov;131(Suppl 6):489-590. doi: 10.1007/s00508-019-01565-0. German. PMID 31792659
- [Background] Blum M, Bachmann K, Wintzer D, Riemer T, Vilser W, Strobel J. Noninvasive measurement of the Bayliss effect in retinal autoregulation. Graefes Arch Clin Exp Ophthalmol. 1999 Apr;237(4):296-300. doi: 10.1007/s004170050236. PMID 10208262
- [Background] Hammer M, Vilser W, Riemer T, Schweitzer D. Retinal vessel oximetry-calibration, compensation for vessel diameter and fundus pigmentation, and reproducibility. J Biomed Opt. 2008 Sep-Oct;13(5):054015. doi: 10.1117/1.2976032. PMID 19021395
- [Background] Marschall S, Sander B, Mogensen M, Jorgensen TM, Andersen PE. Optical coherence tomography-current technology and applications in clinical and biomedical research. Anal Bioanal Chem. 2011 Jul;400(9):2699-720. doi: 10.1007/s00216-011-5008-1. Epub 2011 May 6. PMID 21547430
- [Background] Shiga Y, Asano T, Kunikata H, Nitta F, Sato H, Nakazawa T, Shimura M. Relative flow volume, a novel blood flow index in the human retina derived from laser speckle flowgraphy. Invest Ophthalmol Vis Sci. 2014 May 29;55(6):3899-904. doi: 10.1167/iovs.14-14116. PMID 24876283
- [Background] Werkmeister RM, Schmidl D, Aschinger G, Doblhoff-Dier V, Palkovits S, Wirth M, Garhofer G, Linsenmeier RA, Leitgeb RA, Schmetterer L. Retinal oxygen extraction in humans. Sci Rep. 2015 Oct 27;5:15763. doi: 10.1038/srep15763. PMID 26503332
- [Background] Tian J, Marziliano P, Baskaran M, Tun TA, Aung T. Automatic segmentation of the choroid in enhanced depth imaging optical coherence tomography images. Biomed Opt Express. 2013 Mar 1;4(3):397-411. doi: 10.1364/BOE.4.000397. Epub 2013 Feb 11. PMID 23504041
- [Background] Agrawal R, Gupta P, Tan KA, Cheung CM, Wong TY, Cheng CY. Choroidal vascularity index as a measure of vascular status of the choroid: Measurements in healthy eyes from a population-based study. Sci Rep. 2016 Feb 12;6:21090. doi: 10.1038/srep21090. PMID 26868048
- See also: Description: Medical University of Vienna, Department of Clinical Pharmacology — https://klinische-pharmakologie.meduniwien.ac.at/